CLINICAL TRIAL: NCT02823860
Title: Clinical and Biological Digestive Peritoneal Carcinomatosis Data Base From the French National Network of Peritoneal Surface Malignancies
Acronym: BIG-RENAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL14_0345
Record Dates: First submitted 2016-05-30; First posted 2016-07-06 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Digestive Peritoneal Carcinomatosis
Keywords: Peritoneal carcinomatosis; Biobanking; Biospecimen research; Prospective clinical database; Tissue banking; Quality of Life; various histological subtypes
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Quality of Life; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biospecimens and Quality of Life (QoL) (Other): Only if patient's consent is obtained, biospecimens, including tumor and/or peripheral blood are collected.
  Interventions: Other: Collection of biospecimens and Quality of Life (QoL) assessment

INTERVENTIONS:
Other: Collection of biospecimens and Quality of Life (QoL) assessment — Serum, plasma, buffy coat and formalin-fixed-paraffin-embedded (FFPE). Biospecimens are collected at various stages of diagnostic and therapeutic care.All patients fill out questionnaires of Health related quality of life (QLQ-C30 + QLQ-CR29/STO22, Hospital Anxiety and Depression scale - HAD) and social-demographic survey (Medical Outcome Studies - Social Support Survey- MOS-SSS).

SUMMARY:
To access to good quality biological samples is a prerequisite for high level translational research. The BIG-RENAPE study has been established by the French hyperthermic intraperitoneal chemotherapy centers involved in the management of peritoneal surface malignancies.

The main BIG-RENAPE study aim is to create a large multicentric and prospective repository for biological and tissue samples, which will provide a source of materials for a wide array of health related research studies - BIG-RENAPE Biobank-based research: i) validating known and promising biomarkers; ii) identifying new predictive and prognostic factors; iii) evaluating the impact of current health care strategies; iv) standardizing diagnostic and therapeutic management through guidelines; v) developing new drugs.

The BIG-RENAPE Biobank is certified according to NFS 96-900 as a service of processing, storage and transfer of high quality biological (plasma, serum, buffy coat) and tissue (formalin-fixed-paraffin-embedded) samples. Biospecimens are collected at each stage of diagnostic and therapeutic care. The patient and his derivates are anonymized and registered in a national web database reporting disease status, treatments, surgical procedures, pathological diagnosis, quality of life's assessment and long term follow-up. All participants have given their informed consent before any sample. The BIG-RENAPE study was approved by the local Ethical Committee, based on the assessed compliance to French regulatory rules.

ELIGIBILITY:
Inclusion Criteria:

* Men / women aged over 18 years
* Patients with cancer management and care for peritoneal carcinomatosis of digestive origin
* Patients had histologic/radiologic confirmation of peritoneal disease
* Covered by a Health System where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research;
* Ability of participants to give their informed consent

Exclusion Criteria:

* Minor patient
* Adult unable to consent
* Patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2186 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Resistance to oncological treatments | During the 3-year follow-up
  Resistance to treatments (systemic and intraperitoneal chemotherapy, surgical procedures and targeted therapies) in patients treated for digestive peritoneal carcinomatosis is defined as a change of therapeutic strategy decided during a multidisciplinary meeting.
  The biological and tumoral factors related to resistance of oncological treatments will be identified from the laboratory tests results and histological analyses.
  Biospecimens types: serum, plasma, buffy coat and formalin-fixed-paraffin-embedded (FFPE).
  Biospecimens are collected at various stages of diagnostic and therapeutic care
Presence of biological and tumoral factors related to resistance to oncological treatments | During the 3-year follow-up
  The biological and tumoral factors related to resistance of oncological treatments will be identified from the laboratory tests results and histological analyses.
  Biospecimens types: serum, plasma, buffy coat and formalin-fixed-paraffin-embedded (FFPE).
  Biospecimens are collected at various stages of diagnostic and therapeutic care The biological and tumoral factors related to resistance of oncological treatments will be identified from the laboratory tests results and histological analyses.
  Biospecimens types: serum, plasma, buffy coat and formalin-fixed-paraffin-embedded (FFPE).
  Biospecimens are collected at various stages of diagnostic and therapeutic care

SECONDARY OUTCOMES:
Presence of clinical factors related to resistance to oncological treatments. | During the 3-year follow-up
  Demographic, pathological, clinical information are recorded electronically on a secured Web application and linked to biospecimens identification.
Incidence of recurrence and survival | at 3 years
  Impact of therapeutics strategies on the incidence of recurrence and survival
social characteristics of patients by MOS-SSS test, according to their therapeutic car modalities | at baseline (day 0), 1 month post baseline (M1), 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 months
  The Medical Outcomes Study Social Support Survey (MOS-SSS) is used as a self-administered measure of functional social support for chronically ill persons. The 19 items cover four domains (emotional/informational support, tangible support, positive social interaction, and affection).
quality of life measured by questionnaires (composite measure composed of QLQ-C30, QLQ-CR29 and QLQ-STO22 questionnaires), according to treatment strategies | at baseline (day 0), 1 month post baseline (M1) 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 months
  The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. It incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale.
  The QLQ-CR29 was administered with the QLQ-C30 core questionnaire. It is meant for use among colorectal cancer patients varying in disease stage and treatment modality. The module comprises 29 questions assessing the colorectal cancer-specific symptom scales (disease symptoms, side effects of treatment) and functional scales (body image, sexuality, and future perspective).
  The QLQ-STO22 was administered with the QLQ-C30 core questionnaire. The QLQ-STO22 module contains 22 items regarding dysphagia, pain, reflux, eating restrictions, anxiety, dry mouth, body image, and hair loss.
Intensity of pain perceived by the patient measured by VAS scale | at baseline (day 0), 1 month post baseline (M1), 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 months
  The patient's perception intensity of pain is measured with a Visual Analogue Scale (VAS).
Presence of epidemiological and demographic determinants of delayed access to treatment induction or surgical procedure | During the 3-year follow-up
  Epidemiological and demographic factors will be assessed from the prospective and clinical database.
Presence of prognostic and predictive biomarkers related to resistance to oncological treatments . | During the 3-year follow-up
  The prognostic and predictive biomarkers related to resistance of oncological treatments will be identified from the biological tumoral and clinical data.
behavioral characteristics of patients by HADS Scale, according to their therapeutic car modalities | at baseline (day 0), 1 month post baseline (M1), 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33 and 36 months
  The Hospital Anxiety and Depression Scale (HADS), a self-assessment scale, is used to detect states of depression, anxiety and emotional distress amongst patients who were being treated for a variety of clinical problems.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Glehen, Pr, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud - Service de Chirurgie Générale et Digestive - 165 chemin du grand Revoyet - 69495 Pierre-Bénite, France
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

REFERENCES:
- [Result] Peron J, Mercier F, Tuech JJ, Younan R, Sideris L, Gelli M, Dumont F, Le Roy B, Sgarbura O, Lo Dico R, Bibeau F, Glehen O, Passot G; on behalf BIG-RENAPE working groups. The location of the primary colon cancer has no impact on outcomes in patients undergoing cytoreductive surgery for peritoneal metastasis. Surgery. 2019 Feb;165(2):476-484. doi: 10.1016/j.surg.2018.07.027. Epub 2018 Sep 7. PMID 30197280
- [Result] Bonnefoy I, Mohamed F, Bonnot PE, Benzerdjeb N, Isaac S, Cotte E, Glehen O, Passot G. Risk of Omental Metastases in Patients Undergoing Cytoreductive Surgery for Colorectal Peritoneal Metastases. Dis Colon Rectum. 2020 Sep;63(9):1251-1256. doi: 10.1097/DCR.0000000000001670. PMID 32618618